CLINICAL TRIAL: NCT00643500
Title: Pharmacovigilance Study of Keppra. SPAIN - SKATE : Safety of Keppra as Adjunctive Therapy in Epilepsy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Study Director, UCB
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N01033
Record Dates: First submitted 2008-02-21; First posted 2008-03-26 (Estimated); Last update posted 2013-11-15 (Estimated); Status verified 2009-09

CONDITIONS: Epilepsy, Partial
Keywords: Levetiracetam; Keppra
MeSH Terms: conditions — Epilepsies, Partial | interventions — Levetiracetam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Levetiracetam

SUMMARY:
Patients with partial-onset seizures seen in community-based practices were to be included in this therapeutic use study

* to assess the safety and tolerability of Keppra (Levetiracetam) and to confirm the favorable safety of the drug found during clinical development
* to obtain further information about optimal dosing in daily clinical practice. Compared to previous registration trials, the study population corresponded more closely to that seen in daily clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Male and female older than 16 years;
* Epilepsy with partial onset seizures, with or without secondary generalization;
* At least one concomitant marketed anti-epileptic drug

Exclusion Criteria:

* Safety reasons

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 342 (Actual)
Dates: Start 2002-01; Primary Completion 2003-05 (Actual); Study Completion 2003-05 (Actual)

PRIMARY OUTCOMES:
Adverse event rates, seizure counts and quality of life. | 16 week treatment period

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)